CLINICAL TRIAL: NCT00140257
Title: A Double-Blind, Placebo-Controlled Study of Escitalopram in the Prevention of Depression in Patients With Acute Coronary Syndrome
Brief Title: DECARD: Study of Escitalopram in the Prevention of Depression in Patients With Acute Coronary Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bispebjerg Hospital (Other)
Collaborators: H. Lundbeck A/S (Industry); Danish Heart Foundation (Other); The Danish Medical Research Council (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KF 12-134/04
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2008-12-31 (Estimated); Status verified 2008-12

CONDITIONS: Depression
Keywords: Myocardial Infarction
MeSH Terms: conditions — Depression; Myocardial Infarction | interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Escitalopram

SUMMARY:
Objective: To evaluate the efficacy of preventive treatment with a selective serotonin reuptake inhibitor (SSRI) (escitalopram) in the first year after acute coronary syndromes (ACS).

Methods: 240 patients with acute coronary syndromes (ST-elevation myocardial infarction [STEMI]), non-STEMI or unstable angina) will be enrolled within 8 weeks after ACS and will be randomly assigned to treatment with escitalopram/placebo (5-20 mg) in 52 weeks. Primary outcome measures are the diagnosis of depression and HDS (Hamilton Depression Scale). Psychiatric measurements: SCAN (Schedules for Clinical Assessment in Neuropsychiatry), HDS, HAS (Hamilton Anxiety Rating Scale), Udvalg for Kliniske Undersogelser (UKU) Side Effect Rating Scale, ESSI (Enhancing Recovery in Coronary Heart Disease [ENRICHD] Social Support Instrument), SF-36 (Short Form-36 Health Survey), SCL-92 (Symptom Check List) and BDI (Beck´s Depression Inventory). Cardiological measurements are blood pressure, electrocardiography, echocardiography (left ventricular ejection fraction), heart rate variability and use of medicine.

Discussion: ACS patients with mental illness are usually only diagnosed to a very small extent during admission in a cardiologic department. These patients mainly remain untreated with an increased risk of somatic comorbidity and mortality. Therefore, it is in accordance with ethical principles to conduct a double blind, placebo-controlled study investigating the interface between anxiety, depression and ACS. Even in this blinded study, where one of the groups are treated with placebo, there will be a higher degree of treatment of depressive symptoms due to the low recognition of this problem.

Conclusion: The DECARD study is the first study evaluating the effect of prophylactic treatment of depression in patients with ACS. The study will show if prophylactic treatment will improve cardiac prognosis.

ELIGIBILITY:
Inclusion Criteria:

* ACS
* Randomization within 8 weeks form index hospitalization for ACS
* Age > 18 years
* Not pregnant
* Signed informed consent

Exclusion Criteria:

* Current depression
* Use of antidepressants < 4 weeks
* Previous intolerance to SSRI
* Severe medical conditions
* Severe heart failure
* Alcohol or substance abuse
* Psychosis or dementia
* Current participation in other intervention trials
* Pregnancy and lactation
* Linguistic difficulties

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2004-11; Primary Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Scale
International Classification of Diseases, Revision 10 (ICD-10) Mood Disorder Diagnosis

SECONDARY OUTCOMES:
Cardiac status
Medical comorbidity

CONTACTS AND LOCATIONS:
Overall Officials: Morten Birket-Smith, MD, DMSci, Study Director — Psychiatric Centre Bispebjerg, Bispebjerg University Hospital
Locations (1):
- Bispebjerg University Hospital, Copenhagen, Denmark

REFERENCES:
- [Derived] Hansen BH, Hanash JA, Rasmussen A, Hansen JF, Birket-Smith M. Rationale, design and methodology of a double-blind, randomized, placebo-controlled study of escitalopram in prevention of Depression in Acute Coronary Syndrome (DECARD). Trials. 2009 Apr 7;10:20. doi: 10.1186/1745-6215-10-20. PMID 19351383